CLINICAL TRIAL: NCT01726842
Title: Pediatric Vision Scanner for the Eradication of Amblyopia
Brief Title: Amblyopia and Strabismus Detection Using a Pediatric Vision Scanner
Status: Completed | Type: Observational
Sponsor: Rebiscan, Inc. (Industry)
Collaborators: Retina Foundation of the Southwest (Other)
Responsible Party: Sponsor
Other Study IDs: rebiscan-001
Record Dates: First submitted 2012-10-05; First posted 2012-11-15 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Amblyopia; Strabismus
MeSH Terms: conditions — Amblyopia; Strabismus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Normal Controls: Structurally normal eye with equal visual acuity and normal stereopsis.
  Interventions: Device: Pediatric Vision Scanner
- Referral required: Diagnosed with amblyopia or constant strabismus, categorized based on the GSE.
  Amblyopia:
  * VA <20/40 and 2 logMAR lines difference in normal eye
  * Mild amblyopia (>20/40)
  * Moderate amblyopia (20/40 and <20/100)
  * Severe amblyopia (≥20/100 or worse)
  * Bilateral amblyopia: >4 years age VA<20/40 OU including high hyperopia or high astigmatism.
  Strabismus:
  * Constant: >2 PD at near and or distance.
  * Intermittent: strabismus that could be controlled intermittently either through fusional mechanisms or a compensatory head position.
  Amblyogenic factor categorization:
  * 'Anisometropia'- (1.5 Diopters (D) or more difference in refractive error between the two eyes.
  * 'hypermetropia' (≥3.5 D),
  * 'myopia' (≥-4.0 D),
  * 'astigmatism' (≥1.5 D).
  * 'structural abnormalities' of the eye will not be excluded, but will be considered to have vision loss if visual acuity is 20/40 or worse.
  Interventions: Device: Pediatric Vision Scanner
- Borderline: (no long-term harm to patient if referral is delayed, however the patient does have conditions that might benefit from monitoring): Equal visual acuity and no structural abnormality with any of the following: Amblyogenic factor, intermittent strabismus, structural abnormalities, refractive error, reduced stereopsis.
  Interventions: Device: Pediatric Vision Scanner

INTERVENTIONS:
Device: Pediatric Vision Scanner — Subject is scanned with a 2.5 second pediatric vision scanner device test.

SUMMARY:
The purpose of this project is to compare the performance of the Pediatric Vision Scanner (PVS) with the Gold Standard Examination to determine the effectiveness of the PVS at detecting amblyopia and strabismus.

ELIGIBILITY:
Inclusion:

* 2-6 years old
* complete ophthalmic examination including cycloplegic refraction conducted on the same day or within 3 months
* strabismic, anisometropic, or normal (normal eye examination and refractive error according to AAPOS guidelines)
* parent provides informed consent

Exclusion:

* other ocular disease (includes media opacities, anomalous optic nerve, ptosis, lid hemangioma, conjunctivitis, blepharitis, symptomatic NLD) or systemic disease (JIA, JRA, neurofibromatosis)
* developmental delay
* strabismus surgery in the past 6 months

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children presenting for ophthalmic exam at eye clinic.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2010-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Binocularity score | Day 1

SECONDARY OUTCOMES:
Presence of amblyopia risk factors | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Eileen Birch, PhD, Principal Investigator — Retina Foundation of the Southwest
Locations (1):
- Retina Foundation of the Southwest, Dallas, Texas, United States

REFERENCES:
- [Background] Loudon SE, Rook CA, Nassif DS, Piskun NV, Hunter DG. Rapid, high-accuracy detection of strabismus and amblyopia using the pediatric vision scanner. Invest Ophthalmol Vis Sci. 2011 Jul 7;52(8):5043-8. doi: 10.1167/iovs.11-7503. PMID 21642624